CLINICAL TRIAL: NCT00075868
Title: A Randomized, Double Blind, Placebo-Controlled Phase III Study To Determine The Efficacy Of Sandostatin LAR® Depot (Octreotide Acetate) In Preventing Or Reducing The Severity Of Chemoradiation-Induced Diarrhea In Patients With Anal Or Rectal Cancer
Brief Title: Octreotide in Preventing or Reducing Diarrhea in Patients Receiving Chemoradiotherapy for Anal or Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RTOG-0315; CDR0000349441
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Anal Cancer; Colorectal Cancer; Drug/Agent Toxicity by Tissue/Organ; Radiation Enteritis
Keywords: radiation enteritis; drug/agent toxicity by tissue/organ; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IIIA anal cancer; stage IIIB anal cancer; recurrent anal cancer; stage I anal cancer; stage II anal cancer; recurrent rectal cancer
MeSH Terms: conditions — Anus Neoplasms; Colorectal Neoplasms; Drug-Related Side Effects and Adverse Reactions; Rectal Neoplasms | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sandostatin LAR® Depot (Experimental): Sandostatin LAR® Depot Pre-RT (between day -7 and day -4 of RT) and Day 22 (± 3 days)
  Interventions: Drug: octreotide acetate
- Placebo (Placebo Comparator): Placebo Pre-RT (between day -7 and day -4 of RT) and Day 22 (± 3 days)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: octreotide acetate
  Arms: Sandostatin LAR® Depot
Other: Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Octreotide may be effective in preventing or controlling diarrhea in patients who are undergoing chemoradiotherapy for anal or rectal cancer. It is not yet known whether octreotide is effective in treating diarrhea.

PURPOSE: This randomized phase III trial is studying octreotide in preventing or reducing diarrhea in patients who are undergoing chemoradiotherapy for anal or rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the ability of octreotide to prevent the incidence of moderate, severe, or life-threatening chemoradiotherapy-induced diarrhea (grades 2-4) in patients with anal or rectal cancer.

Secondary

* Compare the quality of life of patients treated with this drug vs placebo.
* Compare the number of hospitalizations and use of antidiarrheal agents (e.g., Imodium®) related to diarrhea (or its complications) in patients treated with these drugs.
* Compare treatment delays and/or dose reductions (chemotherapy and radiotherapy) in patients treated with these drugs.

OUTLINE: This is a double-blind, placebo-controlled, randomized, multicenter study. Patients are stratified according to radiotherapy dose (< 50 Gy vs ≥ 50 Gy), chemotherapy dose (bolus vs continuous), and gender. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive octreotide* intramuscularly (IM) 4-7 days before the start of chemoradiotherapy and on day 22 (± 3 days) during chemoradiotherapy.
* Arm II: Patients receive placebo* IM 4-7 days before the start of chemoradiotherapy and on day 22 (± 3 days) during chemoradiotherapy.

NOTE: *Patients receive a total of 2 injections of octreotide or placebo

In both arms, treatment continues in the absence of unacceptable toxicity.

Quality of life is assessed at baseline, at the completion of chemoradiotherapy, and at 3, 6, 9, and 15 months from the start of chemoradiotherapy.

Patients are followed at 3, 6, 9, and 15 months from the start of chemoradiotherapy.

PROJECTED ACCRUAL: A total of 226 patients (113 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary anal or rectal cancer

  * No metastasis beyond the pelvic regional nodes
* Must be scheduled to receive chemoradiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Liver function tests < 3 times upper limit of normal
* No prior hepatic disease

Renal

* Not specified

Gastrointestinal

* No prior chronic or acute regional enteritis
* No malabsorption syndrome
* No prior inflammatory bowel disease that may exacerbate the radiotherapy toxicity
* No grade 2 or greater uncontrollable diarrhea at baseline
* No prior cholecystitis or gallstones, unless a cholecystectomy has been performed
* No prior incontinence of stool

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled diabetes (e.g., fasting glucose > 250 mg/dL)
* No prior allergy or hypersensitivity to study drug or other related drug or compound
* No other medical condition or mental impairment that would preclude study treatment and compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* Prior chemotherapy allowed

Endocrine therapy

* At least 6 months since prior administration of any of the following:

  * Glucocorticoid therapy
  * Insulin sensitizers (e.g., metformin, pioglitazone, or rosiglitazone)
  * Exogenous growth hormone therapy

Radiotherapy

* See Disease Characteristics
* No prior pelvic radiotherapy
* No prior intensity-modulated radiotherapy
* No concurrent radiotherapy for abdominal cancer
* No concurrent hyperfractionated, split-course, or intensity-modulated radiotherapy
* No brachytherapy prior to or after completion of all external beam radiotherapy

Surgery

* No prior abdominal-perineal resection or other surgical procedure leaving the patient without a functioning rectum
* No colostomy

Other

* More than 30 days since other prior investigational drugs
* No prior octreotide for cancer therapy-related diarrhea
* No concurrent prophylactic antidiarrheal medication

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2003-12; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Prevention of the incidence of moderate, severe, or life-threatening diarrhea

SECONDARY OUTCOMES:
Quality of life
Economic measures
Validity of the Functional Alterations due to Changes in Elimination-Changes in Bowel Function, the Quality of Life-Radiation Therapy Instrument, and the Expand Prostate Index Composite-Bowel questionnaires
Prevention of the incidence of severe or life-threatening (i.e., grade 3-5) diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Babu Zachariah, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Jaffer A. Ajani, MD, Study Chair — M.D. Anderson Cancer Center
Locations (112):
- United States (112):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Saint Agnes Medical Center, Fresno, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Cancer Care Consultants Medical Associates at Daniel Freeman Memorial Hospital, Inglewood, California
  - Leavey Cancer Center at Northridge Hospital Medical Center, Northridge, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Torrance Memorial Medical Center, Torrance, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - St. John's Cancer Center at St. John's Medical Center, Anderson, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Community Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - South Jersey Healthcare Regional Cancer Center, Vineland, New Jersey
  - Long Island College Hospital, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Scott and White Hospital, Temple, Texas
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Columbia St. Mary's Cancer Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - West Allis Memorial Hospital, West Milwaukee, Wisconsin

REFERENCES:
- [Result] Zachariah B, Gwede CK, James J, Ajani J, Chin LJ, Donath D, Rosenthal SA, Kane BL, Rotman M, Berk L, Kachnic LA. Octreotide acetate in prevention of chemoradiation-induced diarrhea in anorectal cancer: randomized RTOG trial 0315. J Natl Cancer Inst. 2010 Apr 21;102(8):547-56. doi: 10.1093/jnci/djq063. Epub 2010 Mar 25. PMID 20339140
- [Result] Zachariah B, James J, Gwede CK, et al.: RTOG 0315: a randomized, double-blind, placebo-controlled phase III study to determine the efficacy of octreotide acetate in preventing or reducing the severity of chemoradiation-induced diarrhea in patients with anal or rectal cancer. [Abstract] J Clin Oncol 25 (Suppl 18): A-4032, 2007.